CLINICAL TRIAL: NCT01371890
Title: Mechanisms and Treatment of Intradialytic Hypertension - Sodium
Acronym: MATCH-Sodium
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 092018-018
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hemodialysis; End-stage Renal Disease; Hypertension; Intradialytic Hypertension
Keywords: hemodialysis; end-stage renal disease; hypertension
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples stored for nitric oxide and endothelin-1 measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intradialytic hypertension: Patients with systolic blood pressure increases > 10 mmHg during 4/6 hemodialysis sessions

SUMMARY:
The purpose of this study is to determine the role of dialysate exposure and fluid removal during hemodialysis in the pathophysiology of intradialytic hypertension.

DETAILED DESCRIPTION:
Specific Aim #1 To determine in a crossover study of 15 maintenance hemodialysis patients with intradialytic hypertension whether standard dialysis with ultrafiltration (dialysate Na of 140), dialysis without ultrafiltration (dialysate Na of 140), or ultrafiltration alone (no dialysate) is associated with the an increase in systolic blood pressure during hemodialysis

Specific Aim #2 To determine in a crossover study of 15 maintenance hemodialysis with intradialytic hypertension whether standard dialysis with ultrafiltration, dialysis without ultrafiltration, or ultrafiltration alone is associated with change in either endothelin-1 or nitric oxide during hemodialysis

SUBSTUDY AIMS

Specific Aim #1 To determine in a randomized 3-week, 2 period crossover study of 15 maintenance hemodialysis patients with intradialytic hypertension whether high vs low dialysate-to-serum Na gradients impairs release of NO, increases ET-1 or causes an acute intradialytic increase in systolic BP,.

Specific Aim #2 TO determine in a randomized 16-week, 2-period crossover study of 30 hemodialysis patients with intradialytic hypertension the effects of 8 weeks of high dialysate-to-plasma Na gradients to 8-weeks of low Na gradients on EC function (FMD and ADMA) and 44 hour ambulatory BP.

ELIGIBILITY:
Inclusion Criteria:

* on hemodialysis > 30 days
* male and female participants, aged 18 to 85 years old, of all races and ethnic origin
* ability to provide informed consent
* Primary nephrologist deems patient is at target dry weight
* KDOQI defined hypertension (predialysis SBP >140 or postdialysis SBP>130) AND
* pre to post hemodialysis SBP increase (>10 mmHg) during 4/6 last HD session

Exclusion Criteria:

* Patients with active cancer or active wounds
* Patient currently on antibiotics or on IV antibiotics within the last month
* BP unable to be measured by routine mechanisms in the upper extremity
* Life expectancy < 6 months
* Inability to provide informed consent
* Larger interdialytic weight gain (>5 kg/treatment on average)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will include up to 45 ESRD patients whose BP increases during hemodialysis. Patients who dialyze at any of the 3 UT Southwestern-affiliated dialysis units will be screened for possible enrollment.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | crossover studies followup 3-16 weeks
  Differences in blood pressure during hemodialysis between treatments

SECONDARY OUTCOMES:
Endothelial cell function | crossover studies with followup of 3-16 weeks
  Differences in nitric oxide and endothelin-1 across treatments Differences in FMD and ADMA between treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jula K Inrig, MD, MHS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern, Dallas, Texas, United States

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822